CLINICAL TRIAL: NCT00967317
Title: Phase III Open Study, Prospective, Multicenter, Randomized, Comparative to the Positive Control for Evaluating the Efficacy and Safety of Auris-Sedina in the Symptomatic Control of Otalgy in Patients With or Without Acute External Otitis.
Acronym: E02OSMAS0108
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratorios Osorio de Moraes Ltda. (Industry)
Responsible Party: Maria Angelina Nardy Mattos, Laboratórios Osório de Moraes Ltda.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E02-OSM-AS-01-08
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2009-08

CONDITIONS: Otitis; Efficacy; Tolerability
Keywords: Auris-Sedina; Otitis; Efficacy; Tolerability
MeSH Terms: conditions — Otitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auris-Sedina (Experimental): Drip 2 drops of the medication with the head tilted and protect with a cotton swab. Repeat the process one at a time until the pain relief. Continue the administration of medication every 3 hours until the pain ceases.
  The medication should be used for a maximum of 3 days when they should return to the doctor.
  Interventions: Drug: Auris-Sedina
- Otosynalar® (Active Comparator): Drip 3 drops in the ear 2 times a day. The medication should be used by more than 3 days after which the patient must return to the doctor.
  Interventions: Drug: Otosynalar®

INTERVENTIONS:
Drug: Auris-Sedina — Drip 2 drops of the medication with the head tilted and protect with a cotton swab. Repeat the process one at a time until the pain relief. Continue the administration of medication every 3 hours until the pain ceases.
  The medication should be used for a maximum of 3 days when they should return to the doctor.
  Arms: Auris-Sedina
Drug: Otosynalar® — Drip 3 drops in the ear 2 times a day. The medication should be used by more than 3 days after which the patient must return to the doctor.
  Arms: Otosynalar®

SUMMARY:
To evaluate the efficacy and tolerability of Auris-Sedina in the symptomatic control of otalgy in patients with and without acute external otitis compared with use of Otosynalar®.

DETAILED DESCRIPTION:
Phase III open Study, multicenter, prospective, randomized entrance of a total of 188 patients, 94 patients will receive medication test and 94 patients will receive Otosynalar®.

Patients will be assessed until the clinical condition has been resolved or a maximum of 3 days.

188 patients of either gender or race, who have at least two of the following symptoms: pain, discharge, tinnitus, ear fullness, subjective hearing loss temporary dizziness or vertigo. And with a clinical or non-acute external otitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with otalgy or not, with acute external otitis ;
* Patients with at least two symptoms of otalgy (pain, discharge, tinnitus, ear fullness, subjective hearing loss temporary dizziness or vertigo) with the Visual Analogic Scale score between 4 and 8 (mild to moderate);
* The patient must present otalgia in one ear;
* Children above 6 years of age;
* Adults over 18 years of age;
* Patients who consent to participate in the study;
* Patients who are female and are of childbearing age should use reliable method of contraception and have negative pregnancy test.

Exclusion Criteria:

* Patients with sensitivity to any component of the formula;
* Patients pregnant or lactating;
* Non visualization of the tympanic membrane of obstruction by cerumen;
* Patients with evidence of any wound or scratch on the ear (ulcerative lesion);
* Patients who are making use of any other medication that might interfere with the evaluation of effectiveness of study (such as antibiotics, antiinflammatory, solutions ear);
* Patients who have severe classification in the Visual Analogic Scale score 9 or 10 in any of the symptoms listed in the questionnaire;
* Patients with otalgy not otological origin;
* Patients with otitis, except acute external otitis ;
* Patients who have epiglottitis;
* The patient with infection;
* Patients who can not follow the procedures clarified in this protocol.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-03 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Visual Analogic Scale, by clinical examination and opinion of the investigator. | 3 days

SECONDARY OUTCOMES:
Of adverse events related to study medication by the Naranjo Algorithm. | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Elie Fiss, Principal Investigator — Faculdade de Medicina do ABC
Locations (1):
- Faculdade de Medicina do ABC, Santo André, São Paulo, Brazil